CLINICAL TRIAL: NCT05562388
Title: Improvement in Nocturia With MAD and Changes in Polysomnographic Value
Brief Title: Mandibular Advancement Device and Changes in Nocturia
Acronym: MAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fernanda Yanez Regonesi (Other)
Collaborators: American Academy of Dental Sleep Medicine (Unknown)
Responsible Party: Sponsor-Investigator, Fernanda Yanez Regonesi, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DENT-22-MAD; 177 - DR - 22 (Other: American Academy of Dental Sleep Mecicine)
Record Dates: First submitted 2022-09-13; First posted 2022-09-30 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-08

CONDITIONS: Obstructive Sleep Apnea; Nocturia; OSA
Keywords: obstructive sleep apnea; oral appliance; nocturia; mandibular advancement device
MeSH Terms: conditions — Sleep Apnea, Obstructive; Nocturia

STUDY DESIGN:
Intervention Model Description: Uncontrolled open label clinical trial. Data gathers from recruitment until appliance delivery will be used allowing each participant to also be their own control, as wait list type of study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- MAD therapy (Experimental): MAD Therapy
  Interventions: Device: Somnodent Classic

INTERVENTIONS:
Device: Somnodent Classic — The efficacy of the device will be evaluated in regards to the response of nocturia. Once patients report an average of voiding per night of less than 2 in the preceding 2 weeks of the follow up they will be classified as responders in term of nocturia and will be evaluated with a second sleep study. Efficacy of MAD will be assessed by comparing the apnea hypopnea index (AHI) values of pre and post sleep study with MAD, and they will be classified as responders if they have 50% improvement in AHI.

SUMMARY:
The main purpose of this study is to test is mandibular advacenment device (MAD) use is associated with reductions in nocturia.

DETAILED DESCRIPTION:
After been informed about the study and informed about risks and benefits, participants will be fitted with a MAD and will be asked to completed questionnaires at baseline, in between follow ups and during follow ups. Nocturia will be assess and appliance will be titrated every 2 weeks until participants report less than 2 voiding per night according to the daily dairies. At that point, second sleep study with MAD in place will be performed to assess treatment effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* English speaker
* >18 y/o
* Obstructive sleep apnea diagnosis with AHI≥5
* ≥ 2 voiding/night at baseline
* Upon clinical examination ≥ 8 teeth per arch, range of mandibular protrusion ≥5 mm
* Consent to participate in the study.

Exclusion Criteria:

* Patients with concomitant diagnosed sleep disorders (i.e. insomnia, narcolepsy, restless legs syndrome, rapid eye movement sleep behavior disorder).
* Prostate/kidney problems (urological disease: (eg overactive bladder, benign prostate hyperplasia)
* Pregnancy
* Heart failure, use of diuretics, diabetes, Parkinson's disease or dementia.
* Patients using combination therapy for the management of obstructive sleep apnea (OSA) (i.e. positive airway pressure (PAP) therapy or positional therapy).
* Upon clinical examination: periodontal disease (>4 mm on periodontal probing, with bleeding on probing, visual signs of periodontal inflammation); tooth horizontal mobility >1 mm, vertical mobility, and unfavorable crown to root ratio; open cavities, loose or fractured restorations, or patient undergoing restorative dental treatments.
* Exaggerated gag reflex.
* Lack of coordination or dexterity.
* Inadequate English comprehension.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2026-03-12 (Estimated); Study Completion 2026-03-12 (Estimated)

PRIMARY OUTCOMES:
To test MAD if associated in changes in nocturia | 15 weeks
  Assessment of efficacy of device in terms of nocturia: Patients will complete daily questionnaires to evaluate voiding at night. Average of 2 preceding weeks of the follow up will be used to determine treatment success in terms of nocturia. Once less than 2 voidings per night is achieved participants will be considers reponders in terms of nocturia and second sleep study will be performed.

SECONDARY OUTCOMES:
Investigate if response to therapy in terms of nocturia is associated with improvement in AHI | 15 weeks
  Once participants report less than 2 voiding per night on average (2 week period), second sleep study will be performed and 50% improvement in apnea hypopnea index will be considered treatment success.

OTHER OUTCOMES:
Changes in quality of life | 15 weeks
  Evaluate changes in quality of life after MAD treatment and see how changes correlate with changes in nocturia. The outcomes will be evaluated with health related quality of life questionnaire at baseline and at the last follow up.
Change in fatigue | 15 weeks
  Evaluate changes in fatigue symptomatology after MAD treatment and see how changes in correlate with changes in nocturia. The outcomes will be evaluated with fatigue assessment scale at baseline and at the last follow up.
Changes in insomnia | 15 weeks
  Evaluate changes insomnia symptomatology after MAD treatment and see how changes correlate with changes in nocturia. The outcomes will be evaluated with insomia severity index questionnaire at baseline and at the last follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Yanez Regonesi, DDS, MS, Principal Investigator — University Of Kentucy
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No